CLINICAL TRIAL: NCT07383649
Title: Initial Safety Lead-in Followed by a Phase II Trial to Study Anti- HCMV Therapy in Breast Cancer Patients With Progressive Intracranial Metastases and CMV Infection (The Breast CMV Study)
Brief Title: Trial to Study Anti- HCMV Therapy in Breast Cancer Patients With Progressive Intracranial Metastases and CMV Infection
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00040888 (HMCC-BR25-001)
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Brain Cancer Metastatic; CMV Viremia
MeSH Terms: conditions — Brain Neoplasms | interventions — Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Anti-HCMV therapy (Oral Valganciclovir) and Standard-of-Care (Experimental): At least 10 patients will be enrolled in the initial safety lead-in followed by the Phase II trial which will include 18 patients. Anti-HCMV therapy, oral Valganciclovir will be given to patients at 900 mg twice a day for 2 weeks. After the induction period, the maintenance will be continued with valganciclovir at 450 mg twice daily for 4 weeks (28 days). CMV PCR, IgG and IgM will be checked at the end of these four weeks. Patients will be followed with physical examinations and assessment of laboratory parameters as required per standard-of-care treatment. Quality-of-life, neurocognitive questionnaires, and MRI brain (if asymptomatic) every 2 months until subsequent intracranial progression or end of study, whichever comes first. Patients will be in follow-up for 24 months.
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir — Valganciclovir inhibits viral DNA polymerase, effectively controlling HCMV reactivation and its associated immunosuppressive effects.
  Dosing for oral Valganciclovir will be based on standard of care dosing as per FDA in patients with HCMV infection. Dose adjustments will be made by the principal investigator for renal function, treatment-related AEs and disease progression according to the manufacturer's recommendations as they are present in individuals and will be assessed on a case-by-case basis.
  Other Names: Valcyte

SUMMARY:
This is a phase II trial with an initial safety lead-in evaluating the efficacy, safety, neurocognitive, and quality-of-life outcomes of anti-cytomegalovirus (CMV) therapy and standard-of-care (SOC) in patients with anti-human cytomegalovirus (HCMV)-reactivated brain metastases. Male and female patients, aged ≥18 years, who have metastatic breast cancer with progressive brain metastases and CMV viremia (> 250 copies/ml) or positive CMV IgG or IgM will be eligible to participate in the trial.

Patients can proceed with SRS as long as at least 1 lesion which is 2 cm or less in a noncritical area in the brain is spared as per the discretion of treating neurosurgeon/radiation oncologist. At least 10 patients will be enrolled in the initial safety lead-in followed by the Phase II trial which will include 18 patients.

Anti-HCMV therapy, oral Valganciclovir will be given to patients at 900 mg twice a day for 2 weeks. After the induction period, the maintenance will be continued with valganciclovir at 450 mg twice daily for 4 weeks (28 days).

DETAILED DESCRIPTION:
This is a phase II trial with an initial safety lead-in evaluating the efficacy, safety, neurocognitive, and quality-of-life outcomes of anti-cytomegalovirus (CMV) therapy and standard-of-care (SOC) in patients with anti-human cytomegalovirus (HCMV)-reactivated brain metastases. Male and female patients, aged ≥18 years, who have metastatic breast cancer with progressive brain metastases and CMV viremia (> 250 copies/ml) or positive CMV IgG or IgM will be eligible to participate in the trial. Patients can proceed with SRS as long as at least 1 lesion which is 2 cm or less in a noncritical area in the brain is spared as per the discretion of treating neurosurgeon/radiation oncologist. Multidisciplinary discussion with neurosurgery and radiation oncology will be needed to determine which patients may be safely enrolled on the trial. At least 10 patients will be enrolled in the initial safety lead-in followed by the Phase II trial which will include 18 patients. The primary endpoint will be to determine the objective response rate after the start of the treatment (anti-HCMV therapy and SOC). Anti-HCMV therapy, oral Valganciclovir will be given to patients at 900 mg twice a day for 2 weeks. Patients will be followed with weekly labs for viral clearance, hematological toxicity, and electrolyte imbalances. CMV PCR, IgG and IgM will be checked at the end of two weeks to monitor for viral clearance. After the induction period, the maintenance will be continued with valganciclovir at 450 mg twice daily for 4 weeks (28 days). Patients will be followed with every 2 weekly labs for hematological toxicity, and electrolyte imbalances. CMV PCR, IgG and IgM will be checked at the end of these four weeks. Pill counting will be done at each follow up to ensure compliance with oral valganciclovir. Patients will be followed with physical examinations and assessment of laboratory parameters as required per standard-of-care treatment. Quality-of-life, neurocognitive questionnaires, and MRI brain (if asymptomatic) every 2 months until subsequent intracranial progression or end of study, whichever comes first. MRI brain will be performed at any symptom onset regardless of study schedule. All MRIs will be evaluated for tumor response and progression using RANO-BM for intracranial and extracranial response using RECIST V1.1.

Patients will be followed for 24 months. Adverse events will be recorded for up to 2 months after treatment discontinuation according to (NCI CTAE) v5. After end of study patients will be followed for survival only.

Correlative studies will include HCMV-DNA copies in serum, and whole-blood based immunophenotyping from baseline to end of anti-CMV treatment. Any craniotomy brain metastatic tissue sample or lumbar puncture done as part of standard of care treatment will also be used for correlative studies. Exploratory blood samples will be transported to Dr Hong Zhao's lab at Fondren building floor 6 in < 4 hours at Room Temperature (RT, 18-25°C) post-collection. Freeze the stabilized blood at -80 °C. The samples will be thawed and lysed using the SmartTube lysis protocol before adding to MDIPA tubes for analysis. Specimens will be stored for up to 3 years after collection. Specimen samples will be accessed by Dr. Hong Zhao's lab for analysis.

Written informed consent is required before performing any trial-specific tests or procedures. Signing of the informed consent form can occur outside the 28-day screening period. All screening evaluations must be completed and reviewed to confirm that patients meet all eligibility criteria before trial entry. Results of standard-of-care tests or examinations performed prior to obtaining informed consent and within 7-28 days prior to trial entry (except where otherwise specified) may be used for screening assessments rather than repeating such tests. The investigator or qualified designer will maintain a screening log to record details of all patients screened and to confirm eligibility or record reasons for screening failure, as applicable.

Neurocognitive testing will consist of the Rey Auditory Verbal Learning Test (RAVLT), Trail Making Test (TMT), and Delis-Kaplan Executive Function System (DKEFS) letter fluency test at baseline and every 8 weeks until end of study or until subsequent intracranial progression, whichever comes first These tests were selected based on the recommendation of the International Cognition and Cancer Task Force (ICCTF). Testing will require approximately 1 hour to complete and will be conducted by the research assistant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged >18 years at the time of consent
2. Breast cancer with progressive brain metastases supra and/or infratentorial. Patients can proceed with SRS as long as at least 1 lesion which is 2 cm or less in a noncritical area in the brain is spared as per the discretion of treating neurosurgeon/radiation oncologist.
3. At least one non irradiated, untreated progressive brain metastases site
4. Serum HCMV DNA by real time PCR > 250 copies/ml or positive CMV Ig G or Ig M.
5. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol. If the patient is unable to consent for any reason a legally authorized guardian may provide consent on their behalf. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act) will be obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
6. Metastatic breast cancer who has systemically no evidence of disease, complete remission, partial remission, stable or progressive disease
7. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
8. Adequate hematology without ongoing transfusion support (hemoglobin > 9 g/dl, absolute neutrophil count (ANC) > 1500 per mm3 , platelets > 100,000 per mm3)
9. Adequate renal and hepatic function (creatinine clearance [CrCL] > 60 mL/min, bilirubin x:≤1.5 upper limit of normal (ULN), aspartate aminotransferase [AST] and alanine aminotransferase [ALT] ≤ 2.5 x ULN and serum albumin ≥ 3 g/dl.
10. Other CMV treatment if clinically indicated per physician's choice
11. Evidence of postmenopausal status or negative serum pregnancy test for premenopausal female patients. Negative serum β-human chorionic gonadotropin pregnancy test within 7 days prior to the first dose of study treatment for premenopausal patients. Women will be considered postmenopausal if they have been amenorrheic for 12 months without an alternative medical cause.

    The following age-specific requirements apply:
12. Women <50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the postmenopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
13. Women ≥50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
14. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up.

Exclusion Criteria:

1. Single resectable intracranial lesion
2. Last intracranial progression free survival > 12 months
3. All progressive brain metastases have been radiated
4. Brain metastases needing immediate local intervention such as mass effect, herniation, active neurological symptoms, increased intracranial pressure, those near vital structures like the motor cortex, proximity to the optic nerve/chiasm or brain stem etc (can still be included if there are any other non-radiated progressive brain metastases) Multidisciplinary discussion with neurosurgery and radiation oncology will be needed to determine which patients may be safely enrolled on the trial.
5. Active pregnancy or breast feeding
6. Women of childbearing potential or fertile men unwilling to use effective contraception (Section 6.2, Table 6) during study and up to three months after treatment discontinuation.
7. Known psychiatric disorder that causes poor cooperation with the trial requirements.
8. Participants with previous other malignancies must have had at least a 3-year disease free interval, except those with non-melanoma skin cancer or carcinoma in situ of cervix
9. Participation in another clinical study with an investigational product within 28 days prior to the first dose of study treatment.
10. Concurrent enrollment in another clinical study unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
11. Unresolved or unstable adverse events (AEs) from prior administration of another investigational drug, per investigators' discretion.
12. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of study treatment.
13. Non-English-speaking subjects will not be enrolled in this study since the neurocognitive tests including DKEFS, RAVLT and TMT are not validated to be scored in other languages.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate with anti-HMCV Therapy and SOC | 6 Weeks
  To estimate the CNS objective response rate (RANO-BM and RECIST V1.1) with anti-HCMV therapy and standard-of-care in metastatic breast cancer patients with progressive brain metastases and CMV viremia or positive CMV IgG or IgM.

SECONDARY OUTCOMES:
Safety and toxicity of anti- HCMV therapy (Valganciclovir) as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTAE) v5 | 16 Weeks
  To assess the safety and toxicity of anti- HCMV therapy (Valganciclovir) in patients with progressive brain metastases and CMV viremia or positive CMV IgG or Ig M, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTAE) v5.
Benefit in median overall survival from start of treatment (anti-HCMV therapy and SOC) until the end of follow up after 24 months or death | 104 Weeks
  To estimate the benefit in median overall survival from start of treatment (anti-HCMV therapy and SOC) until the end of follow up after 24 months or death in patients with treated progressive brain metastases and CMV viremia or positive CMV IgG or IgM.
Prevention of memory decline with anti-HCMV therapy (Valganciclovir) as measured by the mean change in the immediate score on the Rey's Auditory Verbal Learning Test (RAVLT) from baseline to end of study | 104 Weeks
  To estimate the prevention of memory decline with anti-HCMV therapy (Valganciclovir) and SOC in patients with progressive brain metastases and CMV viremia or positive CMV IgG or IgM, as measured by the mean change in the immediate score on the Rey's Auditory Verbal Learning Test (RAVLT) from baseline to end of study
Prevention of memory decline with anti-HCMV therapy (Valganciclovir) and SOC prevention of memory decline with anti-HCMV therapy (Valganciclovir) and SOC | 104 Weeks
  To estimate the prevention of memory decline with anti-HCMV therapy (Valganciclovir) and SOC in patients with progressive brain metastases and CMV viremia or positive CMV IgG or IgM, as measured by the mean change in percent forgetting score on the Rey's Auditory Verbal Learning Test (RAVLT) from baseline to end of study
Prevention of memory decline with anti-HCMV therapy (Valganciclovir) and SOC as measured by the mean change in executive function as measured by Trail Making Test (TMT) from baseline to end of study. | 104 Weeks
  To estimate the prevention of memory decline with anti-HCMV therapy (Valganciclovir) and SOC in patients with progressive brain metastases and CMV viremia or positive CMV IgG or IgM, as measured by the mean change in executive function as measured by Trail Making Test (TMT) from baseline to end of study.
Prevention of memory decline with anti-HCMV therapy (Valganciclovir) and SOC as measured by the mean change in Delis Kaplan Executive Function (DKEFS) Letter Fluency Test from baseline to end of study. | 104 Weeks
  To estimate the prevention of memory decline with anti-HCMV therapy (Valganciclovir) and SOC in patients with progressive brain metastases and CMV viremia or positive CMV IgG or IgM, as measured by the mean change in Delis Kaplan Executive Function (DKEFS) Letter Fluency Test from baseline to end of study.
prevention of quality-of-life decline with anti-HCMV therapy (Valganciclovir) and SOC as measured by the mean change in EORTC QLQ -C30 questionnaire with brain specific module (BN-20) from baseline to end of study. | 104 Weeks
  To estimate the prevention of quality-of-life decline with anti-HCMV therapy (Valganciclovir) and SOC in patients with progressive brain metastases and CMV viremia or positive CMV IgG or IgM, as measured by the mean change in EORTC QLQ -C30 questionnaire with brain specific module (BN-20) from baseline to end of study.
Benefit in post stereotactic radiation progression free survival, defined as time from start of treatment (anti-HCMV therapy and SOC) to subsequent intracranial progression in local radiated site or distant site in the brain | 104 Weeks
  To estimate the benefit in post stereotactic radiation progression free survival, defined as time from start of treatment (anti-HCMV therapy and SOC) to subsequent intracranial progression in local radiated site or distant site in the brain in patients with progressive brain metastases and CMV viremia or positive CMV IgG or IgM.
Median time to distant progression, defined as time from start of treatment (anti-HCMV therapy and SOC) to first sign of distant progression | 104 Weeks
  To determine the median time to distant progression, defined as time from start of treatment (anti-HCMV therapy and SOC) to first sign of distant progression in patients with progressive brain metastases and CMV viremia or positive CMV IgG or IgM.
Systemic objective response rate with anti-HCMV therapy and SOC | 6 Weeks
  To determine the systemic objective response rate with anti-HCMV therapy and SOC in patients with progressive brain metastases and CMV viremia or positive CMV IgG or IgM

OTHER OUTCOMES:
Exploratory Outcome | 104 Weeks
  To evaluate the blood-based correlates of response to anti-HCMV therapy (Valganciclovir) in patients with progressive brain metastases and CMV viremia or positive CMV IgG or IgM. Blood-based correlates of response will include but are not limited to HCMV-DNA copies, and whole-blood based immunophenotyping

CONTACTS AND LOCATIONS:
Overall Officials: Akshjot Puri, M.D., Principal Investigator — The Houston Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Neal Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Taphoorn MJ, Claassens L, Aaronson NK, Coens C, Mauer M, Osoba D, Stupp R, Mirimanoff RO, van den Bent MJ, Bottomley A; EORTC Quality of Life Group, and Brain Cancer, NCIC and Radiotherapy Groups. An international validation study of the EORTC brain cancer module (EORTC QLQ-BN20) for assessing health-related quality of life and symptoms in brain cancer patients. Eur J Cancer. 2010 Apr;46(6):1033-40. doi: 10.1016/j.ejca.2010.01.012. Epub 2010 Feb 22. PMID 20181476
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Shireman JM, White Q, Agrawal N, et al. Genomic Analysis of Human Brain Metastases Treated with Stereotactic Radiosurgery Under the Phase-II Clinical Trial (NCT03398694) Reveals DNA Damage Repair at the Peripheral Tumor Edge. medRxiv [Preprint]. 2023 Apr 24:2023.04.15.23288491. doi: 10.1101/2023.04.15.23288491. PMID: 37131583; PMCID: PMC10153341
- [Background] Berghoff AS, Preusser M. Anti-angiogenic therapies in brain metastases. Memo. 2018;11(1):14-17. doi: 10.1007/s12254-018-0384-2. Epub 2018 Feb 2. PMID 29606977
- [Background] Corroyer-Dulmont A, Valable S, Fantin J, Chatre L, Toutain J, Teulier S, Bazille C, Letissier E, Levallet J, Divoux D, Ibazizene M, Guillouet S, Perrio C, Barre L, Serres S, Sibson NR, Chapon F, Levallet G, Bernaudin M. Multimodal evaluation of hypoxia in brain metastases of lung cancer and interest of hypoxia image-guided radiotherapy. Sci Rep. 2021 May 27;11(1):11239. doi: 10.1038/s41598-021-90662-0. PMID 34045576
- [Background] Voloshin T, Schneiderman RS, Volodin A, Shamir RR, Kaynan N, Zeevi E, Koren L, Klein-Goldberg A, Paz R, Giladi M, Bomzon Z, Weinberg U, Palti Y. Tumor Treating Fields (TTFields) Hinder Cancer Cell Motility through Regulation of Microtubule and Acting Dynamics. Cancers (Basel). 2020 Oct 17;12(10):3016. doi: 10.3390/cancers12103016. PMID 33080774
- [Background] Voloshin T, Kaynan N, Davidi S, Porat Y, Shteingauz A, Schneiderman RS, Zeevi E, Munster M, Blat R, Tempel Brami C, Cahal S, Itzhaki A, Giladi M, Kirson ED, Weinberg U, Kinzel A, Palti Y. Tumor-treating fields (TTFields) induce immunogenic cell death resulting in enhanced antitumor efficacy when combined with anti-PD-1 therapy. Cancer Immunol Immunother. 2020 Jul;69(7):1191-1204. doi: 10.1007/s00262-020-02534-7. Epub 2020 Mar 6. PMID 32144446
- [Background] Kissling C, Di Santo S. Tumor Treating Fields - Behind and Beyond Inhibiting the Cancer Cell Cycle. CNS Neurol Disord Drug Targets. 2020;19(8):599-610. doi: 10.2174/1871527319666200702144749. PMID 32614759
- [Background] Kim EH, Jo Y, Sai S, Park MJ, Kim JY, Kim JS, Lee YJ, Cho JM, Kwak SY, Baek JH, Jeong YK, Song JY, Yoon M, Hwang SG. Tumor-treating fields induce autophagy by blocking the Akt2/miR29b axis in glioblastoma cells. Oncogene. 2019 Sep;38(39):6630-6646. doi: 10.1038/s41388-019-0882-7. Epub 2019 Aug 2. PMID 31375748
- [Background] Chen D, Le SB, Hutchinson TE, Calinescu AA, Sebastian M, Jin D, Liu T, Ghiaseddin A, Rahman M, Tran DD. Tumor Treating Fields dually activate STING and AIM2 inflammasomes to induce adjuvant immunity in glioblastoma. J Clin Invest. 2022 Apr 15;132(8):e149258. doi: 10.1172/JCI149258. PMID 35199647
- [Background] Chen H, Liu R, Liu J, Tang J. Growth inhibition of malignant melanoma by intermediate frequency alternating electric fields, and the underlying mechanisms. J Int Med Res. 2012;40(1):85-94. doi: 10.1177/147323001204000109. PMID 22429348
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225
- [Background] Mehta MP et al. Results from METIS (EF-25), an international, multicenter phase III randomized study evaluating the efficacy and safety of tumor treating fields (TTFields) therapy in NSCLC patients with brain metastases. JCO. 2024; 42, 2008-2008.DOI:10.1200/JCO.2024.42.16_suppl.2008
- [Background] Bokstein F, Blumenthal D, Limon D, Harosh CB, Ram Z, Grossman R. Concurrent Tumor Treating Fields (TTFields) and Radiation Therapy for Newly Diagnosed Glioblastoma: A Prospective Safety and Feasibility Study. Front Oncol. 2020 Apr 21;10:411. doi: 10.3389/fonc.2020.00411. eCollection 2020. PMID 32373508
- [Background] Lu G, Rao M, Zhu P, Liang B, El-Nazer RT, Fonkem E, Bhattacharjee MB, Zhu JJ. Triple-drug Therapy With Bevacizumab, Irinotecan, and Temozolomide Plus Tumor Treating Fields for Recurrent Glioblastoma: A Retrospective Study. Front Neurol. 2019 Jan 31;10:42. doi: 10.3389/fneur.2019.00042. eCollection 2019. PMID 30766509
- [Background] Meletath SK, Pavlick D, Brennan T, Hamilton R, Chmielecki J, Elvin JA, Palma N, Ross JS, Miller VA, Stephens PJ, Snipes G, Rajaram V, Ali SM, Melguizo-Gavilanes I. Personalized Treatment for a Patient With a BRAF V600E Mutation Using Dabrafenib and a Tumor Treatment Fields Device in a High-Grade Glioma Arising From Ganglioglioma. J Natl Compr Canc Netw. 2016 Nov;14(11):1345-1350. doi: 10.6004/jnccn.2016.0145. PMID 27799506
- [Background] Tran DD et al. Final analysis of 2-THE-TOP: A phase 2 study of TTFields (Optune) plus pembrolizumab plus maintenance temozolomide (TMZ) in patients with newly diagnosed glioblastoma. JCO. 2023; 41, 2024-2024.DOI:10.1200/JCO.2023.41.16_suppl.2024